CLINICAL TRIAL: NCT07205952
Title: Automatic Detection of Dyspnea in Mechanically Ventilated, Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: Hospital de Clinicas José de San Martín (Other)
Responsible Party: Principal Investigator, Celica Irrazabal, Director, Intensive Care Unit and Co-Principal Investigator, Hospital de Clinicas José de San Martín
Other Study IDs: 1337-25
Record Dates: First submitted 2025-09-04; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Dyspnea During Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults on invasive mechanical ventilation: Adults of either gender on invasive mechanical ventilation within the preceding 24 hours; and an anticipated need for continued ventilation for ≥24 additional hours. Exclusion criteria are continuous neuromuscular blockade at the time of screening and ventilation using airway pressure release ventilation (APRV).

SUMMARY:
The investigators will conduct a prospective, observational, two-center ICU study of 60 subjects on mechanical ventilation with respiratory failure of any cause.

DETAILED DESCRIPTION:
Inclusion criteria:

* Adults of either sex (≥18 years)
* Non-c0mmunicative, endotracheally intubated in the past 24 hours.
* Expected to require ≥24 hours of mechanical ventilation.

Exclusion criteria:

* Continuous neuromuscular blockade.
* Ventilated on Airway Pressure Release Ventilation mode.

Ventilator measured airway pressure and flow signals will be streamed at 31.25 Hz into 131.1-s time windows (epochs) for up to 5 days. A recursive algorithm will compute individual breath's inspiratory effort (Pmus) and calculate the inspiratory effort time-pressure product (PmusPTP cmH₂O·s·min-¹).

Trained staff will assess the Mechanical Ventilation-Respiratory Distress Observation Scale (MV-RDOS), an intermittent and subjective assessment of dyspnea, at least twice daily. These will be time-matched to the airway signal epochs to determine their degree of correlation by Pearsons R2.

Using receiver operating characteristic (ROC) area under the curve (AUC) analysis, the investigators will determine a dyspnea threshold for PmusPTP equivalent to the dyspnea cut-off for MV-RDOS > 2.6, and report sensitivity/specificity.

To address possible label misclassification, the investigators will train six supervised classifiers on concordant data pairs and apply a unanimity ensemble to label discordant pairs as "dyspneic", not dyspneic" and undetermined". Ensemble determined labels conflicting with those classified by MV-RDOS will be excluded from a secondary analysis.

Primary outcome will be Pearson's R2 (PmusPTP vs MV-RDOS). Secondary outcome will be 28-day ventilator-free days.

ELIGIBILITY:
Inclusion criteria:

* Adults of either sex (≥18 years)
* Endotracheally intubated in the past 24 hours.
* Expected to require ≥24 hours of mechanical ventilation.

Exclusion criteria:

* Continuous neuromuscular blockade.
* Ventilated on Airway Pressure Release Ventilation mode.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults of either sex with respiratory failure of any cause on invasive mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between the pressure-time-product of inspiratory effort and the MV-RDOS score. | One year
  The degree of correlation between the pressure-time-product of inspiratory effort and the MV-RDOS score will be determined with Pearson's coefficient of determination (R2).

SECONDARY OUTCOMES:
Ventilator free days. | One year
  The number of days from the last day of invasive mechanical ventilation to day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Gutierrez, Principal Investigator — The George Washington University School of Medicine and Health Sciences; Celica Irrazabal, MD, Principal Investigator — Hospital de Clínicas José de San Martín
Locations (1):
- Hospital de Clínicas de la Universidad de Buenos Aires, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
1. Excel workbook containing deidentified enrollment information including demographics, mode of ventilation, adverse events during monitoring and outcomes. Also provided will be individual MV-RDOS measurements with time and day after enrollment.
  2. Excel workbook containing paired MV-RDOS measurements and calculated PmusPTP.
  3. Results of machine learning models application to study data.
  4. Program used to develop the machine learning models.
Supporting Information: Study Protocol, SAP
Time Frame: January 1, 2026 through December 31, 2026
Access Criteria: Data are available to qualified investigators on reasonable request by emailing the principal investigator

REFERENCES:
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Gutierrez G. A non-invasive method to monitor respiratory muscle effort during mechanical ventilation. J Clin Monit Comput. 2024 Oct;38(5):1125-1134. doi: 10.1007/s10877-024-01164-z. Epub 2024 May 11. PMID 38733504
- [Background] Gutierrez G. A novel method to calculate compliance and airway resistance in ventilated patients. Intensive Care Med Exp. 2022 Dec 30;10(1):55. doi: 10.1186/s40635-022-00483-2. PMID 36581716
- [Background] Decavele M, Rozenberg E, Nierat MC, Mayaux J, Morawiec E, Morelot-Panzini C, Similowski T, Demoule A, Dres M. Respiratory distress observation scales to predict weaning outcome. Crit Care. 2022 Jun 6;26(1):162. doi: 10.1186/s13054-022-04028-7. PMID 35668459
- [Background] Demoule A, Decavele M, Antonelli M, Camporota L, Abroug F, Adler D, Azoulay E, Basoglu M, Campbell M, Grasselli G, Herridge M, Johnson MJ, Naccache L, Navalesi P, Pelosi P, Schwartzstein R, Williams C, Windisch W, Heunks L, Similowski T. Dyspnoea in acutely ill mechanically ventilated adult patients: an ERS/ESICM statement. Eur Respir J. 2024 Feb 22;63(2):2300347. doi: 10.1183/13993003.00347-2023. Print 2024 Feb. PMID 38387998